CLINICAL TRIAL: NCT05953727
Title: Effects of Low Level Laser Therapy With and Without Proprioceptive Stimulation on Somatosensation, Pain And Gait Parameters in Patients With Discogenic Lumbar Radiculopathy
Brief Title: Low Level LASER Therapy With and Without Proprioceptive Stimulation Among Discogenic Lumbar Radiculopathy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0220
Record Dates: First submitted 2023-06-26; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Lumbar Radiculopathy
Keywords: Discogenic Lumbar Radiculopathy; Gait Parameters; Low-Level Laser Therapy; Numeric pain rating scale
MeSH Terms: conditions — Radiculopathy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy with proprioceptive stimulation (Experimental): Patients will be treated with low level laser therapy and proprioceptive stimulation will also be given.
  Interventions: Other: Low level laser therapy with proprioceptive stimulation
- Low level laser therapy without proprioceptive stimulation (Active Comparator): Patients will be treated with low level laser therapy only.
  Interventions: Other: Low level laser therapy without proprioceptive stimulation

INTERVENTIONS:
Other: Low level laser therapy with proprioceptive stimulation — 10 minutes of low level laser therapy and 10-15 minutes of proprioceptive stimulation and 10 minutes of heating pack. Assessment and data collection will be done at baseline (initial), after 4 weeks of treatment protocol and patients will be followed up for the further 2 weeks to notice and report any change in condition and health status.
  Other Names: Heating packs
  Arms: Low level laser therapy with proprioceptive stimulation
Other: Low level laser therapy without proprioceptive stimulation — 10 minutes of low level laser therapy and 10 minutes of heating pack. Assessment and data collection will be done at baseline (initial), after 4 weeks of treatment protocol and patients will be followed up for the further 2 weeks to notice and report any change in condition and health status.
  Other Names: Heating packs
  Arms: Low level laser therapy without proprioceptive stimulation

SUMMARY:
The aim of this study is to evaluate the effects of low level laser therapy with and without proprioceptive stimulation on somatosensation, pain and gait parameters in patients with discogenic lumbar radiculopathy. The randomized central trial will recruit patients according to convenience sampling into two intervention groups randomly. One group will receive low level laser therapy and proprioceptive stimulation and other group will receive low level laser therapy alone. Heating packs will be given to both groups.

DETAILED DESCRIPTION:
Lumbar disc prolapse occurs when disc material, that is, nucleus pulposus or annulus fibrosis comes out of the intervertebral disc space. The ruptured nucleus interacts with the nearby surrounding nerves, resulting in their compression that in turn causes severe radicular pain. Lumbar disc prolapse is considered as a hallmark of low back pain (LBP). Typically, the pain is distributed bilaterally at the posterior beltline with a sharp, shooting pain running down to the low back, buttocks, and down the thigh along with numbness or tingling sensations. One of the major risk factors for low back pain is lumbar disc prolapse. The prevalence of disc prolapse in lumbar region is 90% (L4-L5 or L5-S1). Low back pain due to disc prolapse is generally self-limiting and of shorter duration

A double blind randomized controlled trial was conducted in 2022 by Ishaq et al. on 110 patients to determine the effectiveness of Low-Level Laser Therapy in Patients with Discogenic Lumbar Radiculopathy and correlation among pain intensity, functional disability, and lumbar range of motion (LROM). The outcomes of the treatment were measured on the first day and then after 18 sessions from each patient's pain intensity, functional disability, L-ROM, and straight leg raise by using visual analogue scale, Oswestry disability index, dual inclinometer, and straight leg raise tests. Experimental group of 55 patients was treated with LLLT and conventional physical therapy while the control group of 55 patients was treated with conventional physical therapy alone. They concluded that LLLT is an efficient adjunct therapy to conventional physical therapy in patients of discogenic lumbar radiculopathy

In the reviewed literature, there seems to be a lack in establishing the effects of low-level laser therapy when combined with proprioceptive stimulation. Discogenic lumbar radiculopathy is very common due to an increased workload, increased number of road traffic accidents, poor postures and socioeconomic status, deficient medical or rehab services, and so on. Thus, there is need to conduct a research to determine the effects of low level laser therapy when combined with proprioceptive stimulation in improving patient's functional status, pain and gait issues.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-70years(27)
* Both male and female patients
* Patients with acute Low Back Pain and unilateral Discogenic Lumbar Radiculopathy with disc bulge confirmed on MRI
* Pain intensity score is 4 or more on the numeric pain rating scale (NPRS)
* Radiating leg pain symptoms for less than 4 weeks
* Numbness and paresthesia in the affected area
* Patients with moderate to severe score (21%-60%) in ODI

Exclusion Criteria:

* Non willing patients
* Patients with severely cognitive disorders
* History of low back pain for more than 4 weeks
* History of any systemic disease such as Stroke, Multiple Sclerosis, Myopathies, Heart Failure etc
* Botulinum toxin injections to any lower extremity muscle in the last 3 months
* Malignancy

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Nottingham Sensory Assessment | 6 weeks
  Multimodal sensory examination includes test of tactile sensation, kinesthesia and stereognosis.
NPRS | 6 weeks
  It is a common pain screening tool use to assess the severity of pain at moment time. It is '0-10' scale where '0' means 'no pain' and '10' means 'worst pain imaginable'.
Step length | 6 weeks
  The distance measured in centimeters between the point of initial contact of one foot and the point of initial contact of the opposite foot is referred to as the step length.
Stride Length | 6 weeks
  The distance covered in centimeters with two consecutive steps, one with each foot.
Walking Cadence | 6 weeks
  Number of steps taken by an individual in one minute

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | 6 weeks
  This is a sub-maximal exercise test used to assess aerobic capacity and endurance. Distance covered over a time of 6 minutes is used to compare changes in performance capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Agile Rehabilitation Complex, Bahawalpur, Punjab Province
  - Bahawal Victoria Hospital, Bahawalpur, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreiner DS, Hwang SW, Easa JE, Resnick DK, Baisden JL, Bess S, Cho CH, DePalma MJ, Dougherty P 2nd, Fernand R, Ghiselli G, Hanna AS, Lamer T, Lisi AJ, Mazanec DJ, Meagher RJ, Nucci RC, Patel RD, Sembrano JN, Sharma AK, Summers JT, Taleghani CK, Tontz WL Jr, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of lumbar disc herniation with radiculopathy. Spine J. 2014 Jan;14(1):180-91. doi: 10.1016/j.spinee.2013.08.003. Epub 2013 Nov 14. PMID 24239490
- [Background] Fardon DF, Williams AL, Dohring EJ, Murtagh FR, Gabriel Rothman SL, Sze GK. Lumbar disc nomenclature: version 2.0: Recommendations of the combined task forces of the North American Spine Society, the American Society of Spine Radiology and the American Society of Neuroradiology. Spine J. 2014 Nov 1;14(11):2525-45. doi: 10.1016/j.spinee.2014.04.022. Epub 2014 Apr 24. PMID 24768732
- [Background] Parker SL, Xu R, McGirt MJ, Witham TF, Long DM, Bydon A. Long-term back pain after a single-level discectomy for radiculopathy: incidence and health care cost analysis. J Neurosurg Spine. 2010 Feb;12(2):178-82. doi: 10.3171/2009.9.SPINE09410. PMID 20121353
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Ahmed I, Bandpei MAM, Gilani SA, Ahmad A, Zaidi F. Effectiveness of Low-Level Laser Therapy in Patients with Discogenic Lumbar Radiculopathy: A Double-Blind Randomized Controlled Trial. J Healthc Eng. 2022 Feb 27;2022:6437523. doi: 10.1155/2022/6437523. eCollection 2022. PMID 35265302
- [Background] Benditz A, Loher M, Boluki D, Grifka J, Vollner F, Renkawitz T, Maderbacher G, Gotz J. Positive medium-term influence of multimodal pain management on socioeconomic factors and health care utilization in patients with lumbar radiculopathy: a prospective study. J Pain Res. 2017 Feb 14;10:389-395. doi: 10.2147/JPR.S128090. eCollection 2017. PMID 28243143
- [Background] National Guideline Centre (UK). Low Back Pain and Sciatica in Over 16s: Assessment and Management. London: National Institute for Health and Care Excellence (NICE); 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK401577/ PMID 27929617